CLINICAL TRIAL: NCT05420909
Title: Overall Survival for Metastatic Colorectal Cancer Patients Matched to CHECKMATE-142
Brief Title: A Study of Overall Survival in Participants With Metastatic Colorectal Cancer (mCRC)
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-7AU
Record Dates: First submitted 2022-06-13; First posted 2022-06-15 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
Keywords: mCRC; Checkmate-142; Nivolumab
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort 1: Participants diagnosed with metastatic colorectal cancer (mCRC) selected from the Flatiron Electronic Health Record database

SUMMARY:
The purpose of this study is to estimate the overall survival (OS) for US participants diagnosed with metastatic colorectal cancer (mCRC) by using Flatiron Health's individual patient level data.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic Colorectal Cancer (CRC) participants in the Flatiron database as defined by:
* Diagnosed with CRC (ICD-9 153.x or 154.x or ICD-10 C18x, or C19x, or C20x, or C21x)
* Pathology consistent with CRC
* At least two documented clinical visits on or after January 1, 2013
* Evidence of Stage IV or recurrent metastatic CRC diagnosed on or after January 1, 2013
* Participants with high levels of microsatellite instability (MSI-H) and/or mismatch repair (MMR) protein deficiency (dMMR)
* Participants who received 2L therapy of interest on or after the initial mCRC diagnosis date
* Participants who had at least 1 month medical data during the prior to and post periods; however, participants who died within 1 month after the index date will not be excluded from the study

Exclusion Criteria:

* Participants <18 years of age at index date
* Participants who received clinical trial drug during the prior or post periods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who were diagnosed with mCRC and received 2L therapy of interest were selected from Flatiron Health's data from January 2013 through March 2019.
  2L therapies of interest included:
  * FOLFIRI and bevacizumab
  * FOLFOX and bevacizumab
  * CAPEOX and bevacizumab
  * FOLFIRI and panitumumab
  * FOLFIRI and ziv-aflibercept
  * FOLFOX, bevacizumab and other (non I-O)
  * FOLFIRI, ziv-aflibercept and other (non I-O)
  * FOLFIRI, bevacizumab and other (non I-O)
  * Nivolumab monotherapy
  * Pembrolizumab monotherapy
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 6 years
Duration of Systemic Treatment | Up to 6 years
  Durations were reported for the first line of therapy prior to the second line (2L) therapy of interest, the 2L therapy of interest, the third line of therapy, and the at least fourth line of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Princeton, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html